CLINICAL TRIAL: NCT05190016
Title: Development of a Multiplex BangasureTM RT-PCR Kit for the Detection of SARS-Corona Virus-2
Brief Title: Efficacy of a Multiplex BangasureTM RT-PCR Kit for the Detection of COVID-19
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: DR. MALA KHAN (Other Government)
Responsible Party: Sponsor-Investigator, DR. MALA KHAN, Director General, Bangladesh Reference Institute of Chemical Measurements (BRICM)
Organization: Bangladesh Reference Institute of Chemical Measurements (BRICM) (Other Government)
Other Study IDs: BANGASURE RT-PCR Kit
Record Dates: First submitted 2022-01-10; First posted 2022-01-13 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cases (Current/fresh): Cases (current/fresh) are defined as those samples which has been tested positive by RT-PCR at IEDCR as a regular screening program and have not been stored in the freezer.
- Cases(stored): Cases (stored) are defined as those samples which has been tested positive by RT-PCR at IEDCR as a regular screening program and have been stored in the -80°C freezer at IEDCR.
- Control (Current/fresh): Control (Current/fresh) are defined as those samples which has been tested negative by RT-PCR at IEDCR as a regular screening program and have not been stored in the freezer.
- Control (stored): Control (stored) are defined as those samples which has been tested negative by RT-PCR at IEDCR as a regular screening program and have been stored in the -80°C freezer at IEDCR

SUMMARY:
The outbreak of the severe acute respiratory syndrome (SARS) corona virus (CoV)-2 continues to increase globally. To control the coronavirus disease 2019 (COVID-19) transmission, diagnose is very important step which would help in the process of quarantine, isolation of the infected person and also in contact tracing. Among the various techniques real-time reverse transcription polymerase chain reaction (rRT-PCR) is mostly used and considers as gold standard method for viral nucleic acid detection as per World Health Organization (WHO) and Centre for Diseases Control (CDC), USA. However, possible false-negative and false-positive results produce misleading consequences, making it necessary to improve existing methods. So, investigators need a robust and reliable PCR kit to detect different kinds of variant of SARS-CoV-2 virus to reduce its transmissibility and take preventive management plan. Beside that to manage the increasing number of testing, investigators are mostly dependent on imported test kit which seems to be very difficult at this pandemic situation and costly. Hence, virulence of SARS-CoV-2 virus may change rapidly due to mutation and country become hot spot so, gene detection RT-PCR kit is time demand. In this point of view, investigator's aim to develop an validate multiplex rRT-PCR qualitative diagnostic method, which targets two viral genes E (envelope protein), N (nucleocapsid gene, according to the CDC, USA guidelines for the development of RT-PCR kit and one human gene RNase P as internal control simultaneously.

This is a case control study where will analyze 120 samples (60 COVID-19 positive and 60 COVID-19 negative both fresh and frozen) from Institute of Epidemiology, Disease Control and Research (IEDCR). This specimen will be blinded before supplying over to NILMRC/Contact ROL/ Bangladesh Clinical Trail Limited (BCTL), Dhaka, Bangladesh for Bangladesh Reference Institute for Chemical Measurements (BRiCM) RT-PCR Kit. Required in house validation will also be conducted as per International Council for Harmonization (ICH) and FDA guideline and also external validation will be carried in different Director General of Health Service (DGHS), Bangladesh approved COVID-19 diagnostic laboratory. Data will be analyzed by computer using Statistical Package for the Social Sciences (SPSS) software and will be presented into the frequency table, graph and chart according to the requirements.

DETAILED DESCRIPTION:
Introduction:

The corona virus COVID-19 pandemic is the defining global health crisis of our time and the greatest challenge that have faced since World War Two. The pandemic is much more than a health crisis; it's also an unprecedented socio-economic crisis. Since its identification in the region of Wuhan, China, not only the virus has spread across 213 countries/territories with 209 million cases and 4.39 million globally but also could put 400million people out of their jobs as The International Labor Organization estimates.

To contain the spread of disease, multidisciplinary strategies have been launched in different regions of the world, including implementing social distancing, maintaining personal hygiene, contact tracing, and implementing quarantine, travel restrictions, and lock downs. A widely accepted method is testing for SARS-CoV-2, typically utilizing nasopharyngeal swab specimens. Patients tested positive require appropriate clinical management by either effective isolation or quarantine at home for mild symptoms or within health care facilities for moderate to severe symptoms. In addition, wide-scale testing provides more informative epidemiologic data for drafting policies on disease monitoring and control. Many approaches have been proposed to detect SARS-CoV-2 virus in nasopharyngeal fluids such as multiplex RT-PCR, CRISPR/Cas12, and CRISPR-Cas3, lateral flow immunoassay, paper-based bimolecular sensors, SHERLOCK testing in one pot, DNA aptamer, loop-mediated isothermal amplification (LAMP), etc. Among these methods, nucleic acid amplification-based tests are the most common for the diagnosis of SARS-CoV-2.

In addition, US CDC suggest a protocol for the detection of SARS-CoV-2, based on the amplification of two regions of the nucleocapsid gene, namely N1and N2, and a human internal control gene RNase P (RP). In addition to these strategies, efforts to develop SARS-CoV-2 detection methods with high efficiency and accuracy, with less reaction time and effort, are still ongoing.

However, despite being considered as the gold standard for SARS CoV-2 detection, testing has lagged behind in many countries because of various factors, most important being supply chain issues with lack of reagents and adequate test kits. Therefore, many patients (both symptomatic and asymptomatic) remain untested and hence are potentially contributing to community spread of the virus.

If Bangladesh can produce its own RT-PCR kits which is no less in quality in terms of sensitivity, specificity etc. than that would mitigate the shortage of RT-PCR kit as investigators are totally dependent on imported test kits and also save foreign currency. Moreover, RT-PCR test kits are very temperature sensitive and need to maintain the cold chain for its quality which can be mitigated by developing local RT PCR kit. Additionally, many variant of SARS-CoV-2 has been developed due to mutation, which has shown more virulence and high transmission rate. So, development of new RT PCR kit which can detect newer strain can be extremely helpful.

So, here investigator's aim to develop the three gene detectable robust RT-PCR kit that will be country first and give reliable result of different kinds of variant of SARS-CoV-2 virus for reducing its transmissibility and taking preventive management plan 2. Objectives of the Study:

1. General Objectives: Primary objectives are aimed to develop multiplex real-time reverse transcription polymerase chain reaction (rRT-PCR) to detect of SARS-CoV-2.
2. Secondary Objectives: For the best RT-PCR performance, the combination of E and N gene targets should be optimized.

   3. Methodology: 3.1. Study type & purpose: This is a case control and observational study in which two existing groups frozen and fresh samples are identified and compared.

   3.2. Place of study:
   * Institute Epidemiology Disease Control and Research (IEDCR)
   * M/S. Clinical Research Organization Ltd 3.3. Sample Collection Site(s):
   * Institute Epidemiology Disease Control and Research (IEDCR) or
   * National Institute of Laboratory Medicine & Referral Centre (NILMRC), Dhaka, Bangladesh.

   3.4. Duration of study: • 3 months (November, 2021 to January, 2022) after getting Ethical Clearance from Bangladesh Medical Research Council.

   3.5. Study Population/sample selection 3.5.1 CRO will receive testing samples from IEDCR. IEDCR and BCTL/CROL as CRO have memorandum of understanding (MoU) for different collaborative research work. So, NILMRC/ BCTL/CROL will receive a total 120 sample from IEDCR for the evaluation of RT-PCR kit efficiency. Of the 120 samples, 60 will be stored samples (30 COVID-19 known positive and 30 COVID-19 negative samples) which have been kept at -80°C lab freezers at IEDCR facilities and another 60 fresh specimens (30 COVID-19 positive and 30 COVID-19 negative samples) which are being tested at IEDCR. Samples with discordant results will be rejected before testing by BRiCM RT PCR kit. That is, more than 120 identified samples from IEDCR might be needed to analyze by imported RT-PCR kits and extraction kit at BCTL/CROL. This is how 120 samples will be selected for performance evaluation of BRiCM RT-PCR kit.

   3.5.2 To avoid biasedness and conflicts of interest, sponsor and PI/co-investigators will be blinded to the sample ID and positive/negative status of the samples and clinical records of the patients. The positive/negative status of both stored and fresh samples will be identified at IEDCR before sending to BCTL/CROL. That is, BCTL/CROL personnel will also be blinded to sample identity document (ID) and positive negative/negative status before analysis. Finally, the CRO head will send the performance evaluation certificate to the PI or Sponsor.

   3.5.3. Statistical Basis of Sample Size:

   Formulae:

   The study is conducted on 120 participants (60 stored known positive & negative and 60 fresh known positive & negative). To achieve desire absolute accuracy (n) in estimating efficiency of RT-PCR the minimum sample size estimated following following the Discrete Bernoulli Probability Function as follows:

   Alfa= 5% D= absolute Accuracy (%) with 95% confidence. Desired Absolute accuracy n D Alfa=5% Z=1.96 10 30.99% n D= (1.96)/(2* Square Root (SQRT) (n)) 20 21.91% 100 9.80% 30 17.89% 120 8.94% 100 9.80% 200 6.93% 300 5.66% 400 4.90% 1000 3.10% 10000 0.98% 20000 0.69% 30000 0.57% 100000 0.3% 3.6 Sample Selection Criteria 3.6.1 Inclusion criteria: Samples with Positives RT-PCR results with Ct value≤35 for the COVID-19 genes at IEDCR will be selected as COVID-19 positive. Samples with negative RT-PCR results with no amplification for the COVID-19 genes at IEDCR will be selected as COVID-19.
   * Gender: All
   * Age: 5 to 70 years (Child, Adult, Older Adult) 7.8.2. Exclusion criteria
   * Samples with equivocal/ambiguous RT-PCR results in terms of sigmoidal curve and Ct value will be excluded.

   Consents from the patients are not required because the CRO will receive the specimens from IEDCR as per MOU with IEDCR. So there is no requirement of patient's enrollment and consents and CRF from the CRO side.

   3.7 Data Collection Procedure: COVID-19 positive samples will be confirmed by laboratory findings of positive RT-PCR results for the viral RNA.

   3.8 Data Analysis: The sensitivity, specificity, positive predictive value and negative predictive value of BRiCM COVID-19 real time RT-PCR kit will be determined. The chi-square test (two sided) will be performed for comparing categorical variables. A p value of ≤0.05 will be considered as the level of significant association. Alongside sensitivity, specificity, positive predictive value and negative predictive value, Kappa coefficient, positive likelihood ratio, and negative likelihood ratio will also be calculated.

   3.9 The database is safeguarded against unauthorized access by established security procedures; appropriate backup copies of the database and related software files shall be maintained. Databases are backed up by the database administrator in conjunction with any updates or changes to the database.

   3.10 The Investigator must make study data accessible to the monitor and authorized representatives. The Investigator must provide interim study report with data at every three months interval to the principle investigator. As per requirement study report and data may be provided to Bangladesh Medical Research Council (BMRC) and Directorate General of Drug Administration (DGDA). The Investigator must ensure the reliability and availability of source documents.

   3.11 Monitoring visits will be conducted by principle investigator, co- investigator as well as the representatives according to Guidelines for Good Clinical Practice (GCP).

   3.12 In order to maintain subject confidentiality, only a site number, subject number and subject initials will identify all study subjects on Case Records Forms (CRF) and other documentation submitted to the investigator. Additional subject confidentiality issues (if applicable) are covered in the Clinical Study Agreement.

   3.13 All records will be kept secret to the PI, co-investigators, sponsor except IEDCR responsible persons who are in charge. Samples will be identified as code/ID number and date at IEDCR before sending to BCTL/Contact Research Organization Limited (CROL) 4. For this study the mentioned institute IEDCR/Bangladesh Clinical Trail Limited (BTCL)/CRO Ltd. has the capability to conduct the clinical trial to find out the efficacy of kit through their existing resource. Beside that CRO can manage the chemical, reagent and technology if any needed for the study as per MoU between funding agencies.

   5. Conflict of the interest BRiCM is the funding agency of proposed COVID-19 RT-PCR kit, is a statutory body functioning under the administrative control of the Ministry of Science and Technology. It is a research organization and a reference institute in the area of chemical measurements. It is neither a commercial enterprise nor a profit making organization. According to constitutional sanction the principal responsibility of BRiCM is to carry on research leading to such innovation that will add value to the government effort for ensuring welfare of the people.

ELIGIBILITY:
Inclusion Criteria:

* Samples with Positives RT-PCR results with Ct value≤35 for the COVID-19 genes at IEDCR will be selected as COVID-19 positive.
* Samples with negative RT-PCR results with no amplification for the COVID-19 genes at IEDCR will be selected as COVID-19.

Exclusion Criteria:

* Samples with equivocal/ambiguous RT-PCR results in terms of sigmoidal curve and Ct value will be excluded.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: IEDCR and BCTL/CROL as CRO have MoU for different collaborative research work. So, NILMRC/ BCTL/CROL will receive a total 120 sample from IEDCR for the evaluation of RT-PCR kit efficiency. Of the 120 samples, 60 will be stored samples (30 COVID-19 known positive and 30 COVID19 negative samples) which have been kept at -80°C lab freezers at IEDCR facilities and another 60 fresh specimens (30 COVID-19 positive and 30 COVID19 negative samples) which are being tested at IEDCR. Samples with discordant results will be rejected before testing by BRiCM RT PCR kit. That is, more than 120 identified samples from IEDCR might be needed to analyze by imported RT-PCR kits and extraction kit at BCTL/CROL. This is how 120 samples will be selected for performance evaluation of BRiCM RT-PCR kit.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Performance evaluation of BRiCM COVID-19 RT-PCR | 1 month
  Determine Performance evaluation of BRiCM COVID-19 RT-PCR with extracted viral RNA by using standard viral RNA extraction kit for the detection of SARS-CoV-2 virus in nasopharyngeal swab specimens collected in the nationwide COVID-19 screening program. RNA extraction from fresh Nasopharyngeal Swab sample in the Viral Transport Medium (VTM) of COVID-19 patients from IEDCR (30 positive and 30 negative) Analysis of COVID-19 RNA samples using RT-PCR.

SECONDARY OUTCOMES:
Reduce the price and enhance the efficiency to detect COVID-19 by BRiCM COVID-19 RT-PCR kit | 1 month
  Supply locally manufacturer COVID-19 reverse transcription polymerase chain reaction (RT-PCR) kit to govt. and private hospitals for diagnosis of COVID-19 patients. RNA extraction from frozen nasopharyngeal swab sample in viral transport medium (VTM) of COVID-19 patients from IEDCR (30 positive and 30 negative) analysis of COVID-19 RNA samples using reverse transcription polymerase chain reaction (RT-PCR).

CONTACTS AND LOCATIONS:
Overall Officials: MAMUDUL HASAN RAZU, MSc, Principal Investigator — Scientific Officer; MD MONIRUZZAMAN, BSc, Study Chair — Senior Scientific Officer; PRANAB KARMAKER, Dr, Study Chair — Senior Scientific Officer; ZABED BIN AHMED, MSc, Study Chair — Senior Scientific Officer; MD IQBAL HOSSAIN, MSc, Study Chair — Scientific Officer; MD FAZLE ALAM RABBI, Dr, Study Chair — Lecturer
Locations (1):
- Institute for Developing Science and Health Initiatives, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) is not applicable for this study because the study will analyze frozen/fresh specimens from IEDCR. IEDCR will receive these samples as the Reference Laboratory for COVID-19 sample analysis from different hospitals, clinics, trial and testing booths. IEDCR also receives samples for validation from COVID-19 laboratory across the country. So, there will be no subject enrollment and no requirement of IPD. Hence, IPD sharing plan is not applicable in this regard.

REFERENCES:
- [Background] Bedford J, Enria D, Giesecke J, Heymann DL, Ihekweazu C, Kobinger G, Lane HC, Memish Z, Oh MD, Sall AA, Schuchat A, Ungchusak K, Wieler LH; WHO Strategic and Technical Advisory Group for Infectious Hazards. COVID-19: towards controlling of a pandemic. Lancet. 2020 Mar 28;395(10229):1015-1018. doi: 10.1016/S0140-6736(20)30673-5. Epub 2020 Mar 17. No abstract available. PMID 32197103
- [Background] Choi S, Ki M. Estimating the reproductive number and the outbreak size of COVID-19 in Korea. Epidemiol Health. 2020;42:e2020011. doi: 10.4178/epih.e2020011. Epub 2020 Mar 12. PMID 32164053
- [Background] Ulloa S, Bravo C, Parra B, Ramirez E, Acevedo A, Fasce R, Fernandez J. A simple method for SARS-CoV-2 detection by rRT-PCR without the use of a commercial RNA extraction kit. J Virol Methods. 2020 Nov;285:113960. doi: 10.1016/j.jviromet.2020.113960. Epub 2020 Aug 22. PMID 32835738
- [Background] Kudo E, Israelow B, Vogels CBF, Lu P, Wyllie AL, Tokuyama M, Venkataraman A, Brackney DE, Ott IM, Petrone ME, Earnest R, Lapidus S, Muenker MC, Moore AJ, Casanovas-Massana A; Yale IMPACT Research Team; Omer SB, Dela Cruz CS, Farhadian SF, Ko AI, Grubaugh ND, Iwasaki A. Detection of SARS-CoV-2 RNA by multiplex RT-qPCR. PLoS Biol. 2020 Oct 7;18(10):e3000867. doi: 10.1371/journal.pbio.3000867. eCollection 2020 Oct. PMID 33027248
- [Background] Broughton JP, Deng X, Yu G, Fasching CL, Servellita V, Singh J, Miao X, Streithorst JA, Granados A, Sotomayor-Gonzalez A, Zorn K, Gopez A, Hsu E, Gu W, Miller S, Pan CY, Guevara H, Wadford DA, Chen JS, Chiu CY. CRISPR-Cas12-based detection of SARS-CoV-2. Nat Biotechnol. 2020 Jul;38(7):870-874. doi: 10.1038/s41587-020-0513-4. Epub 2020 Apr 16. PMID 32300245
- [Background] Ali Z, Aman R, Mahas A, Rao GS, Tehseen M, Marsic T, Salunke R, Subudhi AK, Hala SM, Hamdan SM, Pain A, Alofi FS, Alsomali A, Hashem AM, Khogeer A, Almontashiri NAM, Abedalthagafi M, Hassan N, Mahfouz MM. iSCAN: An RT-LAMP-coupled CRISPR-Cas12 module for rapid, sensitive detection of SARS-CoV-2. Virus Res. 2020 Oct 15;288:198129. doi: 10.1016/j.virusres.2020.198129. Epub 2020 Aug 18. PMID 32822689
- [Background] Chen Z, Zhang Z, Zhai X, Li Y, Lin L, Zhao H, Bian L, Li P, Yu L, Wu Y, Lin G. Rapid and Sensitive Detection of anti-SARS-CoV-2 IgG, Using Lanthanide-Doped Nanoparticles-Based Lateral Flow Immunoassay. Anal Chem. 2020 May 19;92(10):7226-7231. doi: 10.1021/acs.analchem.0c00784. Epub 2020 May 5. PMID 32323974
- [Background] Joung J, Ladha A, Saito M, Kim NG, Woolley AE, Segel M, Barretto RPJ, Ranu A, Macrae RK, Faure G, Ioannidi EI, Krajeski RN, Bruneau R, Huang MW, Yu XG, Li JZ, Walker BD, Hung DT, Greninger AL, Jerome KR, Gootenberg JS, Abudayyeh OO, Zhang F. Detection of SARS-CoV-2 with SHERLOCK One-Pot Testing. N Engl J Med. 2020 Oct 8;383(15):1492-1494. doi: 10.1056/NEJMc2026172. Epub 2020 Sep 16. No abstract available. PMID 32937062
- [Background] Chen Z, Wu Q, Chen J, Ni X, Dai J. A DNA Aptamer Based Method for Detection of SARS-CoV-2 Nucleocapsid Protein. Virol Sin. 2020 Jun;35(3):351-354. doi: 10.1007/s12250-020-00236-z. Epub 2020 May 25. No abstract available. PMID 32451881
- [Background] Zhen W, Berry GJ. Development of a New Multiplex Real-Time RT-PCR Assay for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Detection. J Mol Diagn. 2020 Dec;22(12):1367-1372. doi: 10.1016/j.jmoldx.2020.09.004. Epub 2020 Sep 19. PMID 32961315
- [Background] Khan S, Tombuloglu H, Hassanein SE, Rehman S, Bozkurt A, Cevik E, Abdel-Ghany S, Nabi G, Ali A, Sabit H. Coronavirus diseases 2019: Current biological situation and potential therapeutic perspective. Eur J Pharmacol. 2020 Nov 5;886:173447. doi: 10.1016/j.ejphar.2020.173447. Epub 2020 Aug 5. PMID 32763302
- [Background] Yan C, Cui J, Huang L, Du B, Chen L, Xue G, Li S, Zhang W, Zhao L, Sun Y, Yao H, Li N, Zhao H, Feng Y, Liu S, Zhang Q, Liu D, Yuan J. Rapid and visual detection of 2019 novel coronavirus (SARS-CoV-2) by a reverse transcription loop-mediated isothermal amplification assay. Clin Microbiol Infect. 2020 Jun;26(6):773-779. doi: 10.1016/j.cmi.2020.04.001. Epub 2020 Apr 8. PMID 32276116
- [Background] Moran A, Beavis KG, Matushek SM, Ciaglia C, Francois N, Tesic V, Love N. Detection of SARS-CoV-2 by Use of the Cepheid Xpert Xpress SARS-CoV-2 and Roche cobas SARS-CoV-2 Assays. J Clin Microbiol. 2020 Jul 23;58(8):e00772-20. doi: 10.1128/JCM.00772-20. Print 2020 Jul 23. No abstract available. PMID 32303565
- [Background] Landis JR, Koch GG. The measurement of observer agreement for categorical data. Biometrics. 1977 Mar;33(1):159-74. PMID 843571